CLINICAL TRIAL: NCT02016469
Title: A Randomized, Controlled, Single-blind Study of Effects of Pectin on Flora Intestinal Colonization and Maintenance After Fecal Transplantation to Patients With Inflammatory Bowel Disease
Brief Title: Effects of Pectin on Flora Intestinal Colonization and Maintenance After Fecal Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, weiyao, doctor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBDBP-1
Record Dates: First submitted 2013-12-10; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Pectins; Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- co-transplantation of FMT and pectin (Experimental): 300ml Bacterial suspension (from 60g fresh stool )given for the first day and 20g pectin given from the second to the sixth day for total five days
  Interventions: Other: co-transplantation of FMT and pectin
- single fecal microbiota transplantation (Active Comparator): 300ml Bacterial suspension (from 60g fresh stool )given for the first day
  Interventions: Other: single fecal microbiota transplantation
- give pectin 20g/d (Active Comparator): pure give pectin 20g/d for five days
  Interventions: Dietary Supplement: pure give pectin 20g/d for five days

INTERVENTIONS:
Other: co-transplantation of FMT and pectin — 300ml Bacterial suspension (from 60g fresh stool )for fecal microbiota transplantation the first day and 20g pectin given continuously for total five days
  Arms: co-transplantation of FMT and pectin
Other: single fecal microbiota transplantation — single fecal microbiota transplantation once the first day
  Arms: single fecal microbiota transplantation
Dietary Supplement: pure give pectin 20g/d for five days — pure give pectin 20g/d for five days
  Arms: give pectin 20g/d

SUMMARY:
The purpose of this study is to evaluate the effect and safety of pectin and fecal microbiota transplantation on patients with inflammatory bowel disease. The investigators hypothesize that patients who take pectin can promote the migration of probiotics in intestine engraftment, reduce pathogenic agents'adhesion to intestinal mucosa, cut down the inflammation, and to maintain intestinal flora diversity and steady state in a long time.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic relapsing disease, including ulcerative colitis (UC) and Crohn's disease (CD). Although the etiology of IBD is unknown, but more and more evidence show that the inappropriate immune response to intestinal commensal bacteria leading to dysbiosis, and pathogens further act to the mucosal lymphoid tissue, causing IBD. Has yet not to determine the specific one or more pathogens as the cause of IBD,but literatures confirm the changes of diversity of the intestine flora.Based on the current awareness of changes in the intestinal flora in IBD, fecal microbiota transplantation (FMT) proposed in recent years to rebuild the intestine flora balance to achieve therapeutic purposes. But fecal bacteria of patients can not consistent with donor's for a long term after transplantation and therefore it is not an ideal way for disease control. Maintaining the diversity of flora in a long time so that well controlled the disease become the breakthrough of fecal microbiota transplantation in the treatment of inflammatory bowel disease.

Pectin is a soluble dietary fiber (DF), produced by the gut flora after a series of fermentation with many metabolites such as short chain fatty acids (SCFA) which supply the energy for epithelial cells, regulate intestinal PH and intestinal motility and join effort in immune regulation with intestinal lymphoid tissue. Previous studies showed that: water-soluble dietary fiber with the action of intestinal flora can cut the inflammatory cytokines, prevent inflammation and induce regulatory T cells, but the type and dose of dietary fiber used were different in different studies, and no studies have confirmed whether dietary fiber could adjusted the flora colonization ability in patients with IBD. We conceive that pectin by some mechanism to promote the migration of probiotics in intestine engraftment, reduce pathogenic agents' adhesion of intestinal mucosa, cut inflammation, and to maintain intestinal flora diversity and steady state in a long time, and than achieve the goal of continue to ease IBD.

ELIGIBILITY:
Inclusion Criteria:

for UC

1. Patients should be in the age range of 18 - 70 years;
2. Patients should have clinical, imaging, endoscopic and histological diagnosis of UC;
3. Patients should have a UCDAI score of more than 2 and less than 10 or stage at S1/S2 in Montreal Rank at enrollment;
4. Patients receiving a stable dose of concomitant medication (aminosalicylates, oral corticosteroids) for at least 4 weeks are eligible;
5. Patients are capable of providing written informed consent and obtained at the time of enrollment;
6. Patients are willing to adhere to the study visit schedule and other protocol requirements.

for CD:

1. Patients should be in the age range of 18 - 40 years;
2. Patients should have clinical, imaging, endoscopic and histological diagnosis of early CD*;
3. Patients should have a CDAI score of more than 150 and less than 400and have a C-reactive protein (CRP) level of more than10mg/L at enrollment;
4. Patients receiving a stable dose of concomitant medication (aminosalicylates, oral corticosteroids) for at least 4 weeks are eligible;
5. Patients are capable of providing written informed consent and obtained at the time of enrollment;
6. Patients are willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Women who are pregnant or lactating at the time of enrollment, or who intend to be during the study period
2. Patients may confuse the findings or there exist any other additional risk history
3. Patients with end-stage disease or is expected likely to die during the study
4. Patients are participating in other clinical trials or participated within 3 months prior to transplantation
5. Outbreaks, infectious (viruses, bacteria, parasites, or other microorganisms) colitis, scheduled for abdominal surgery,take probiotics / prebiotics / synbiotics / antibiotic / PPI (past 1 month) orally, severe anemia (Hbg <6g/dl), heart cerebrovascular accident, bypass, stent implantation surgery in the last 6 months, coagulation disorders, immune suppression status (defined as: immunosuppressive drugs, a history of opportunistic infections within one year recurrent ,oral ulcers, multiple lymphadenopathy, neutropenia, etc.), major abdominal transplant surgery in the last 3 months, have took TNF-α monoclonal antibody 2 month before transplantation or planned to take within one month after transplantation, a history of megacolon -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
diversity and steady state of the stool | 6 months
  Change from Baseline in diversity and steady state of the stool every week within one month after the intervention and three and six months after intervention

SECONDARY OUTCOMES:
Erythrocyte sedimentation rate | 6 months
  Change from Baseline in ESR 1st,3st,6st month after intervention
C-reactive protein | 6 months
  Change from Baseline in CRP 1st,3st,6st month after intervention
Fecal calcium protein | 6 months
  Change from Baseline in Fecal calcium protein 1st,3st,6st month after intervention
Adverse reactions after fecal microbiota transplantation and/or take pectin | 1 week
  every day within one week after the intervention
Crohn's disease activity index | 6 months
  Change from Baseline in CDAI two weeks,one,three and six months after intervention
Ulcerative Colitis disease activity index | 6 months
  Change from Baseline in UCDAItwo weeks,one,three and six months after intervention
the simple endoscopic score for CD | 6 months
  Change from Baseline in SEC-CD 3st,6st months after intervention
Ulcerative Colitis endoscopic index of severity | 6 months
  Change from Baseline in UCDEIS 3st and 6st month after intervention
diversity and steady state of the Intestinal mucosa | 6 months
  Change from Baseline in diversity and steady state of the intestinal mucosa three and six months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Jinling hosptal,Medical School of Nanjing University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Ge X, Ding C, Gong J, Tian H, Wei Y, Chen Q, Gu L, Li N. [Short-term efficacy on fecal microbiota transplantation combined with soluble dietary fiber and probiotics in the treatment of slow transit constipation]. Zhonghua Wei Chang Wai Ke Za Zhi. 2016 Dec 25;19(12):1355-1359. Chinese. PMID 28000190
- [Derived] Wei Y, Gong J, Zhu W, Tian H, Ding C, Gu L, Li N, Li J. Pectin enhances the effect of fecal microbiota transplantation in ulcerative colitis by delaying the loss of diversity of gut flora. BMC Microbiol. 2016 Nov 3;16(1):255. doi: 10.1186/s12866-016-0869-2. PMID 27809778